CLINICAL TRIAL: NCT06576154
Title: The Role of Antibiotic Prophylaxis in Lowering Wound Infection Rates Post-Open Repair of Primary Elective Groin Hernias in High-Risk Patients: A Randomized Control Trial.
Brief Title: The Role of Antibiotic Prophylaxis in Lowering Wound Infection Rates Post-Open Repair of Primary Elective Groin Hernias in High-Risk Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Aleppo (Other)
Collaborators: Aleppo University Hospital Resident Team (Unknown)
Responsible Party: Principal Investigator, Ahmad Yamen Arnaout, Principal Investigator, University of Aleppo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AP-GH-OE-2023-HR
Record Dates: First submitted 2024-08-21; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Antibiotic Prophylaxis; Wound Infection; Groin Hernia
Keywords: Groin hernia; Postoperative complications; Wound infection; Surgical site infection; High-risk patients
MeSH Terms: conditions — Wound Infection; Hernia, Inguinal; Postoperative Complications; Surgical Wound Infection | interventions — Cefazolin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prophylaxis antibiotics Group (Experimental): Patients with Antibiotic Prophylaxis post-open Repair of Primary Elective Groin Hernias in High-Risk Patients.
  Interventions: Drug: Cefazolin 1000 MG
- Non-antibiotics Group (No Intervention): Patients without Antibiotic Prophylaxis post-open Repair of Primary Elective Groin Hernias in High-Risk Patients.

INTERVENTIONS:
Drug: Cefazolin 1000 MG — * Medication: Cefazolin
  * Dosage: 1 gram
  * Administration Timing: A single dose will be administered preoperatively.
  Arms: Prophylaxis antibiotics Group

SUMMARY:
This study aims to investigate the impact of antibiotic prophylaxis on reducing wound infection rates following open repair of primary elective groin hernias in high-risk patients.

DETAILED DESCRIPTION:
This study will be a randomized controlled trial involving high-risk patients undergoing open repair of primary elective groin hernias. Participants will be randomized into two groups: one receiving antibiotic prophylaxis and the other serving as the control group. The study will assess the incidence of wound infections postoperatively in both groups to determine the effectiveness of antibiotic prophylaxis in lowering infection rates.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the study.
* Elderly patients aged over 60 years.
* Patients with Diabetes.
* Or obese patients with a BMI greater than 35.
* Or immunocompromised patients.
* Or American Society of Anesthesiologists (ASA) physical status classification 2 or more, with a history of more than 10 years.

Exclusion Criteria:

* Non-cooperative patients for regular follow-up.
* Therapeutic Indication for.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Overall Complication Rate | up to 30 days after the surgery.
  Overall complication rate; graded by the Clavien- Dindo complications classification system
Wound infection/ Surgical site infection | up to 30 days after the surgery.
  has been defined and classified as superficial incisional, deep incisional, and organ/ space_ surgical site infection by the Centers for Disease Control and Prevention (CDC) (Anderson 2014; Ban 2017; Berríos-Torres 2017).

SECONDARY OUTCOMES:
Mortality Rate | up to 30 days after the surgery.
  The measure of the number of deaths at the end of the study.
Hospital stay | up to 30 days after the surgery.
  In days: Number of days, patient in hospital since admission.

OTHER OUTCOMES:
Other Adverse events | up to 30 days after the surgery.
  Any adverse events will be observed during the follow-up period.

CONTACTS AND LOCATIONS:
Locations (1):
- Aleppo University Hospital, Aleppo, Syria

IPD SHARING:
Plan to Share IPD: No